CLINICAL TRIAL: NCT06096090
Title: A Phase II Clinical Trial of Interleukin-2 (IL-2) in Patients With Mild to Moderate Alzheimer's Disease
Brief Title: Phase II Clinical Trial of Interleukin-2 in AD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Alireza Faridar, Assistant Professor, The Methodist Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO00030798
Record Dates: First submitted 2023-10-17; First posted 2023-10-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Interleukin-2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Aldesleukin every 4 weeks (Active Comparator)
  Interventions: Drug: Interleukin-2
- Aldesleukin every 2 weeks (Active Comparator)
  Interventions: Drug: Interleukin-2
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Interleukin-2 — Low dose Interleukin-2 (Aldesleukin) administration to expand Regulatory T cells
  Arms: Aldesleukin every 2 weeks; Aldesleukin every 4 weeks
Drug: Placebo — Placebo administration
  Arms: Placebo

SUMMARY:
Neuroinflammation is a significant component of Alzheimer disease (AD). Our group recently demonstrated that regulatory T cells (Tregs) have a compromised phenotype and reduced suppressive function in AD patients, skewing the immune system toward a proinflammatory status and potentially contributing to disease progression. Low dose interleukin-2 (IL-2) is now viewed as a promising immunoregulatory drug with the capacity to selectively expand and restore functional Tregs. This study is a phase II, randomized, double-blind, placebo-controlled study to assess low dose IL-2 therapy in AD patients. Up to 40 Alzheimer's disease patients in the mild- to moderate clinical dementia stages (MMSE scores: 12-26) will be randomized to five-day-courses of subcutaneous IL-2 or placebo for a total of 6 months. We will evaluate the safety and tolerability of IL-2 treatment and the possible effects of IL-2 treatment on peripheral and central inflammation. The expected time participants will be in the study is 30 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of probable Alzheimer disease according to National Institute on Aging-Alzheimer's Association (NIA-AA) criteria
2. Male or female age 50 to 86 years
3. MMSE between 12-26
4. Total bilirubin less than or equal to 1.5mg/dL
5. Alanine aminotransferase level (ALT) and aspartate aminotransferase (AST) less than or equal to two times normal,
6. Albumin greater than or equal to 3.0mg/dL
7. Serum creatinine less than or equal to 1.5 mg/dL
8. White Blood Count (WBC) >3,500/mm3; platelets >100,000/mm3; hematocrit (HCT) >32%.
9. INR<1.4 If on medications affecting cognition (rivastigmine, galantamine, donepezil, memantine), participants must be on stable dosage for at least 4 weeks prior to screening and should remain at a stable dosage during the course of the study.
10. English language speaking
11. Formal education of eight or more years
12. Stable pharmacological treatment of any other chronic conditions for at least 30 days prior to screening

Exclusion Criteria:

1. Serious, active bacterial, fungal or viral infection, active or latent tuberculosis
2. History of severe pulmonary dysfunction
3. Severe cardiac dysfunction defined as left ventricular ejection fraction <40% if an echocardiogram is medically indicated to clarify ongoing symptoms or EKG findings.; a history of non-controlled cardiac arrhythmias; history of cardiac tamponade; Unstable angina or MI in the last 3 months
4. Hypersensitivity or allergy to IL-2
5. History of bowel ischemia/perforation, or GI bleeding requiring surgery
6. Hospitalization or change of chronic concomitant medication within one month prior to screening.
7. History of hemorrhage or infarct or > 3 lacunar infarcts, cerebral contusion, encephalomalacia, aneurysm, vascular malformation, subdural hematoma, hydrocephalus, space-occupying lesion (e.g. abscess or brain tumor with the exception of small incidental meningiomas) in prior CT or MRI.
8. Clinical or laboratory findings consistent with:

   1. Other primary degenerative dementia, (dementia with Lewy bodies, fronto-temporal dementia, Huntington's disease, Jacob-Creutzfeld Disease, Down's syndrome, etc.)
   2. Other neurodegenerative condition (Parkinson's disease, amyotrophic lateral sclerosis, etc.)
   3. Seizure disorder
   4. History of infectious, metabolic or systemic diseases affecting the central nervous system (syphilis, vitamin B12 or folate deficiency, other laboratory values, etc.)
   5. Clinically significant abnormal T4 or TSH
9. A current DSM-V diagnosis of active major depression, schizophrenia or bipolar disorder. Patients with depressive symptoms successfully managed by a stable dose of an antidepressant are allowed entry.
10. Clinically significant, advanced or unstable disease that may interfere with outcome evaluations, such as:

    1. Respiratory insufficiency
    2. Bradycardia (<45/min.) or tachycardia (>100/min.)
    3. Poorly managed hypertension (systolic >160 mm Hg and/or diastolic >95 mm Hg) or hypotension (systolic <90 mm Hg and/or diastolic <60 mm Hg)
    4. Uncontrolled diabetes defined by HbA1c >8%
11. History of cancer within 3 years of screening with the exception of fully excised non-melanoma skin cancers or non-metastatic prostate cancer that has been stable for at least 6 months.
12. History of acute/chronic hepatitis B or C and/or carriers of hepatitis B
13. Disability that may prevent the patient from completing all study requirements (e.g. blindness, deafness, severe language difficulty, etc.).
14. Within 4 weeks of screening visit or during the course of the study, concurrent treatment with antipsychotic agents (except risperidone ≤1.5 mg/day, quetiapine ≤100 mg/day, olanzapine ≤5 mg/day, and aripiprazole ≤10 mg/day), antiepileptics (except lamotrigine, gabapentin and pregabalin for nonseizure indications), centrally active anti-hypertensive drugs (e.g., clonidine, l-methyl dopa, guanidine, guanfacine, etc.), opiate analgesics, systemic corticosteroids, psychostimulants, antiparkinsonian medications (except for non-parkinsonian indications) and mood stabilizers (e.g., valproate, lithium), sedatives, and anxiolytics with the exception that use of short- to medium-acting benzodiazepines for treatment of insomnia is permitted, however, use of sedatives or hypnotics should be avoided for 8 hours before administration of cognitive tests.
15. Nootropic drugs except stable AD meds (acetylcholinesterase inhibitors and memantine.
16. Suspected or known drug or alcohol abuse, i.e. more than approximately 60 g alcohol (approximately 1 liter of beer or 0.5 liter of wine) indicated by elevated MCV significantly above normal value at screening
17. Suspected or known allergy to any components of the study treatments.
18. Intake of investigational drug within the previous 30 days or five half-lives of the investigational drug, whichever is longer.
19. Exposure to passive immunotherapies for AD (e.g. monoclonal antibodies) within the previous 180 days to dosing, and BACE inhibitors within the previous 30 days to dosing.
20. Chronic steroid or interferon therapy
21. Contraindication to undergoing an LP including, but not limited to: inability to tolerate an appropriately flexed position for the time necessary to perform an LP; INR >1.4 or other coagulopathy; platelet count of <100,000/μL; infection at the desired lumbar puncture site; taking anti-coagulant medication within 90 days of screening (Note: low dose aspirin is permitted); suspected non-communicating hydrocephalus or intracranial mass; prior history of spinal mass or trauma.
22. Any condition, which in the opinion of the investigator makes the patient unsuitable for inclusion.

Ages: 50 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and the tolerability of IL-2 in AD patients | 6 months treatment phase
  Primary endpoint:
  - Number of participants with adverse events and with abnormal laboratory findings (serum chemistry, hematology)

SECONDARY OUTCOMES:
To investigate the impact of IL-2 administration on the blood Treg population in AD patients | 6 months treatment phase
  Secondary Endpoint:
  - Change in Treg percentage out of total CD4 cells

CONTACTS AND LOCATIONS:
Locations (1):
- Houston Methodist Research Institute, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Faridar A, Gamez N, Li D, Wang Y, Boradia R, Thome AD, Zhao W, Beers DR, Thonhoff JR, Nakawah MO, Roman GC, Volpi JJ, Toledo JB, George M, Davis CS, Pascual B, Grundman M, Masdeu JC, Appel SH. Low-dose interleukin-2 in patients with mild to moderate Alzheimer's disease: a randomized clinical trial. Alzheimers Res Ther. 2025 Jul 4;17(1):146. doi: 10.1186/s13195-025-01791-x. PMID 40615880